CLINICAL TRIAL: NCT02273622
Title: Nutritional Intervention Study to Evaluate the Effect of Hydroxytyrosol on Phase II Enzymes in Healthy Subjects
Brief Title: Human Study of Hydroxytyrosol on Phase II Enzymes in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IMDEA Food (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IMD PI011
Record Dates: First submitted 2014-10-15; First posted 2014-10-24 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
Keywords: hydroxytyrosol; dietary supplement; gene expression regulation
MeSH Terms: interventions — 3,4-dihydroxyphenylethanol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- hydroxytyrosol 5 mg (Experimental): each participant will alternately by the three arms of the study (hydroxytyrosol 5 mg and 20 mg and placebo
  Interventions: Dietary Supplement: hydroxytyrosol
- hydroxytyrosol 20 mg (Experimental): each participant will alternately by the three arms of the study (hydroxytyrosol 5 mg and 20 mg and placebo
  Interventions: Dietary Supplement: hydroxytyrosol
- placebo (Placebo Comparator): each participant will alternately by the three arms of the study (hydroxytyrosol 5 mg and 20 mg and placebo
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: hydroxytyrosol — Pilot study with 20 participants, each participant will alternately by the two arms of the study (hydroxytyrosol 5 mg and 20 mg) and control, during 6 weeks.
  Arms: hydroxytyrosol 20 mg; hydroxytyrosol 5 mg
Dietary Supplement: placebo
  Arms: placebo

SUMMARY:
Explore the detoxifying potential of hydroxytyrosol and its effects on Phase II enzyme expression (leading to xenobiotics detoxification in the liver).

DETAILED DESCRIPTION:
Hydroxytyrosol is peculiar to olives (and, hence, to olive oil) and is being exploited as a potential supplement or preservative to be employed in the nutraceutical, cosmeceutical, and food industry. One of the properties described for the hydroxytyrosol is its high antioxidant activity. Also, hydroxytyrosol is able to modulate several enzymatic activities linked to cardiovascular disease. Animal experiments confirm hydroxytyrosol retains its antioxidant activity once ingested (though the human metabolic pathway has been elucidated and shows extensive glucuronidation and subsequent urinary excretion), protects from second hand smoke-induced oxidative damage, inhibits platelet aggregation, ameliorates lipid profile and decreases atherosclerosis development, increases brain cell resistance to oxidation and mitochondrial membrane potential Several mechanisms have been proposed to explain how biologically polyphenols protect against degenerative diseases. It is now thought more likely that some phytochemicals, including polyphenols, are processed by the body as xenobiotics. They stimulate stress- related cell signalling pathways that result in increased expression of genes encoding cytoprotective genes. Nrf2 (NF-E2-related factor 2) is a transcription factor which binds to the Antioxidant Response Element (ARE) in cells and thus regulates enzymes involved in antioxidant functions or detoxification (e.g. thioredoxin reductase-1 and glutathione peroxidases). Polyphenols might increase gene transcription of Nrf2 mediated by such response elements. This provides grounds for the theory of hormesis, i.e. when mild stress triggers defense mechanisms. In the case of polyphenols it indicates how they could have an indirect antioxidant action.

That is why plans to carry this study to explore the detoxifying potential of hydroxytyrosol and its effects on Phase II enzyme expression (leading to xenobiotics detoxification in the liver). It´ll be a randomized crossover, pilot study examining the effects of two doses of hydroxytyrosol, in the form of a commercially-available raw mixture: 1) providing 5 mg/d; 2) 25 mg/d, for one week with a one-week washout period in between, during 6 weeks.

The investigators will recruit 20 healthy volunteers, from within those who participate in the Genyal Platform studies AT IMDEA-Food Institute.

ELIGIBILITY:
Inclusion Criteria:

* Male gender with age range 20-40 years
* Signed patient informed consent

Exclusion Criteria:

* BMI < 19 and >26
* Subjects with a diagnosis of diabetes mellitus, dyslipidemia, hypertension and other cardiometabolic diseases.
* Subjects with dementia, mental illness or diminished cognitive function.
* Subjects with serious diseases (hepatic, renal, cardiovascular, etc.)
* Subjects who refuse to make the 24 hour urine collection and blood samples under study.
* Subjects with allergy or intolerance to olive and derivatives.
* Subjects with drug treatment of any kind.
* Current smoking.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-10; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Detoxifying potential of hydroxytyrosol and its effects on Phase II enzyme expression (leading to xenobiotics detoxification in the liver). | Change of Baseline and after one week hydroxytyrosol and placebo administration
  The analyses of gene expression will be carried out at the ad-hoc platform in use at IMDEA-Food (see www.food.imdea.org for details). Total RNA will be extracted from mononuclear cells with TRI Reagent (Sigma-Aldrich, Inc., St. Louis, MO, USA) and purified with RNeasy MiniElute Cleanup Kit (Qiagen, Hilden, Germany). Recovered RNA will be quantified using a Nanodrop ND-1000 v3.5.2 spectrophotometer (Nanodrop TechnologyR, Cambridge, UK). RNA integrity will be assessed using 1.6% agarose gel, 1× TBE. RNA will be judged suitable for array hybridization only if samples exhibited intact bands corresponding to 18S and 28S ribosomal RNAs. During the study blood samples will be obtained from venous puncture and blood samples will be collected in tubes containing EDTA, maintained on ice and rapidly centrifuged to obtain plasma. Plasma will be immediately distributed in aliquots for the different determinations and stored at -70 °C until analysis.

SECONDARY OUTCOMES:
Number of participants with change in different anthropometrics parameters | Change of Baseline and after one week hydroxytyrosol and placebo administration
  The different anthropometrics parameters are: weight, height, body mass index, fat mass, lean mass
Number of participants with change in different biochemical parameters | Change of Baseline and after one week hydroxytyrosol and placebo administration
  The different biochemical parameters are: Lipid profile (TG, CT, LDL-C, HDL-C), oxidation (LDL-ox, 8-iso PGF2α), inflammatory (PCRu, TNFα, IL1β, VCAM1, ICAM; TXB2).
Concentration of hydroxytyrosol and metabolites in urine | Change of Baseline and after one week hydroxytyrosol and placebo administration
  Urine sampling will be performed before administration of the substance (t=0) and after 24 h post dose. Urinary HT and metabolites will be measured by mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Visioli, Prof, Principal Investigator — IMDEA Food
Locations (1):
- IMDEA-Food, Madrid, Madrid, Spain

REFERENCES:
- [Background] Visioli F, Galli C, Plasmati E, Viappiani S, Hernandez A, Colombo C, Sala A. Olive phenol hydroxytyrosol prevents passive smoking-induced oxidative stress. Circulation. 2000 Oct 31;102(18):2169-71. doi: 10.1161/01.cir.102.18.2169. PMID 11056087
- [Background] Visioli F, Galli C, Bornet F, Mattei A, Patelli R, Galli G, Caruso D. Olive oil phenolics are dose-dependently absorbed in humans. FEBS Lett. 2000 Feb 25;468(2-3):159-60. doi: 10.1016/s0014-5793(00)01216-3. PMID 10692578
- [Background] Visioli F, Caruso D, Plasmati E, Patelli R, Mulinacci N, Romani A, Galli G, Galli C. Hydroxytyrosol, as a component of olive mill waste water, is dose- dependently absorbed and increases the antioxidant capacity of rat plasma. Free Radic Res. 2001 Mar;34(3):301-5. doi: 10.1080/10715760100300271. PMID 11264904
- [Background] Visioli F, Bellosta S, Galli C. Oleuropein, the bitter principle of olives, enhances nitric oxide production by mouse macrophages. Life Sci. 1998;62(6):541-6. doi: 10.1016/s0024-3205(97)01150-8. PMID 9464466
- [Derived] Crespo MC, Tome-Carneiro J, Burgos-Ramos E, Loria Kohen V, Espinosa MI, Herranz J, Visioli F. One-week administration of hydroxytyrosol to humans does not activate Phase II enzymes. Pharmacol Res. 2015 May-Jun;95-96:132-7. doi: 10.1016/j.phrs.2015.03.018. Epub 2015 Mar 30. PMID 25836918